CLINICAL TRIAL: NCT00241280
Title: Study Intended to Evaluate the Safety and Effectiveness of a Johnson & Johnson Vision Care Inc, (JJVCI) Contact Lens for Use on an Extended-wear Basis for up to 7 Days (6 Nights).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CR-1480
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Control (Active Comparator): etafilcon A contact lens being worn 7 days/6 nights.
  Interventions: Device: etafilcon A
- Test (Experimental): galyfilcon A contact lens being worn 7 days/6 nights.
  Interventions: Device: galyfilcon A

INTERVENTIONS:
Device: etafilcon A
  Arms: Control
Device: galyfilcon A
  Arms: Test

SUMMARY:
Study in the US intended to evaluate the safety and effectiveness of a Johnson & Johnson Vision Care Inc, (JJVCI) contact lens for use on an extended-wear basis for up to 7 days (6 nights).

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 18 years of age.
* The subject must read and sign the statement of informed consent and be provided with a copy of the form.
* Minimum of 7 days of successful lens wear
* Contact lens prescription requiring between -1.00 to -6.00 D spherical power
* Less than 1.00 D of astigmatism in either eye

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2005-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Steven S. Grant, OD, Costa Mesa, California
  - Cole, Cole, and Krohn, Fresno, California
  - Fukai and Associates, Louisville, Colorado
  - Peter C. Donshik, MD, Bloomfield, Connecticut
  - Dr. Ted Brink and Associates, Jacksonville, Florida
  - Jack J. Yager, OD, Orlando, Florida
  - Clayton Eye Center, Morrow, Georgia
  - Eyecare Associates, Bloomington, Illinois
  - Drs. Hawks, Besler & Rogers, Gardner, Kansas
  - Lee Rigel, East Lansing, Michigan
  - Univ Missouri at St. Louis, College of Optometry, St Louis, Missouri
  - InSight Eyecare, Warrensburg, Missouri
  - Drs. Quinn, Quinn and Associates, Athens, Ohio
  - Central Ohio Eyecare, Columbus, Ohio
  - Kenji Hamada, OD, Grants Pass, Oregon
  - West Hills Vision Center, Moon Township, Pennsylvania
  - Kenneth A. Young, OD, Brentwood, Tennessee
  - Gary W. Jerkins, MD, Nashville, Tennessee
  - Premier Vision, Amarillo, Texas
  - Charles Wegman, OD, Carrollton, Texas
  - Wishnow-Sugar Vision Group, Katy, Texas
  - First Eye Care Plano, Plano, Texas
  - Dr. William Bogus, Salt Lake City, Utah
  - Scott Jens, OD, Middleton, Wisconsin
  - Snowy Range Vision Center, Laramie, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 504 Subjects were enrolled in this study. 1 subject did not meet the eligibility. 2 subjects were randomized to the control lens group, but were not dispensed lenses. 247 subjects were randomized to the Control lens and 254 subjects were randomized to the Test lens.
Groups:
- Control: Etafilcon A: Subjects that were randomly assigned to wear Control lens.
- Test: Galyfilcon A: Subjects that were randomly assigned to wear the Test lens.
Period: Overall Study
Arm/Group | Control: Etafilcon A | Test: Galyfilcon A
Started | 247 | 254
Completed | 199 | 186
Not Completed | 48 | 68
Not completed — Adverse Event | 2 | 6
Not completed — Discomfort | 11 | 16
Not completed — Pregnancy | 1 | 5
Not completed — Lost to Follow-up | 5 | 8
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Protocol Violation | 4 | 10
Not completed — Relocation | 4 | 4
Not completed — Unsatisfactory Physiological Response | 1 | 1
Not completed — Unsatisfactory Visual Response | 1 | 1
Not completed — Diabetic | 1 | 0
Not completed — Subject Ineligible/Dispensed | 9 | 6
Not completed — Dispensed incorrect test article | 1 | 2
Not completed — Unacceptable Fit | 0 | 1
Not completed — Scheduling Conflict | 0 | 2
Not completed — History of Ocular Surgery | 0 | 1
Not completed — Coating on Lens | 1 | 0
Not completed — Excessive Dryness | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline population consists of subjects that were randomized to receive either the Test or Control lens.
Groups:
- Control: Etafilcon A: Subjects that were randomized to receive the Control lens etafilcon A
- Test: Galyfilcon A: Subjects that were randomized to receive the Test lens galyfilcon A
- Total: Total of all reporting groups
Arm/Group | Control: Etafilcon A | Test: Galyfilcon A | Total
Number analyzed (Participants) | 247 | 254 | 501
Age, Continuous [Mean (Full Range); unit: years] | 31.7 [18 to 51] | 32.8 [18 to 60] | 32.2 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 172 | 322
  Male | 97 | 82 | 179
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 11 | 10 | 21
  White | 203 | 217 | 420
  African-American | 16 | 13 | 29
  Hispanic | 12 | 13 | 25
  Asian-Indian | 1 | 1 | 2
  Other | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 247 | 254 | 501

OUTCOME MEASURES:

1. Primary Outcome: Monocular Contact Lens Snellen Visual Acuity Worse Than 20/40
Description: Percentage of subject eyes reported with visual acuity worse than 20/40 at each study visit.
Time Frame: Follow-up Visits- 24 hr, 1, 4, 12, 24,36, and 52 weeks
Population: The analysis population consists of subjects that completed all study visits, without a major protocol deviation. The analysis was conducted on these subject eyes.
Measure: Number; unit: Percentage of Subjects Eyes
Units Other Than Participants: Eyes
Groups:
- Control: Etafilcon A: Subjects that were randomly assigned to wear the Control lens.
- Test: Galyfilcon A: Subjects that were randomly assigned to wear the Test lens.
  It was reported that for one subject eye, that the contact lens was dirty during the visual acuity testing.
Arm/Group | Control: Etafilcon A | Test: Galyfilcon A
Number analyzed (Participants) | 199 | 186
Number analyzed (Eyes) | 398 | 372
Percentage of Subjects Eyes
  24-Hr. Follow-up, N=396, 370 | 0 | 0
  1-week Follow-up, N=393, 366 | 0 | 0
  4-week Follow-up, N=392, 370 | 0 | 0
  12-week Follow-up, N=388, 370 | 0 | 0
  24-week Follow-up, N=390, 370 | 0 | .27
  36-week Follow-up, N=390 , 365 | 0 | 0
  52-week Follow-up, N=390, 368 | 0 | 0

2. Primary Outcome: Rate of Contact Lens Related Serious and Significant Events (SSE)
Description: The number of Contact-Lens related Serious and Significant Adverse Events were reported for each study lens. The incidence of rates of contact-lens related SSEs were calculated as (# of subjects that experienced an event)/(total # subjects). If there were multiple diagnostic findings, the event was categorized under the highest event level diagnostic.
Time Frame: Throughout the duration of the study (1 Year)
Population: All subjects that were dispensed a study lens.
Measure: Number; unit: percentage of Subjects
Arm/Group | Control: Etafilcon A | Test: Galyfilcon A
Number analyzed (Participants) | 247 | 254
percentage of Subjects | 2.4 | 5.9

ADVERSE EVENTS:
Time Frame: Throughout the duration of the Study (1 Year)
Groups:
- Test: Galyfilcon A: Subjects that were randomly assigned to wear Test lens.
Arm/Group | Control: Etafilcon A | Test: Galyfilcon A
Serious Adverse Events (participants affected / at risk) | 0/247 | 1/254
Other Adverse Events (participants affected / at risk) | 23/247 | 43/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: Etafilcon A (N=247) | Test: Galyfilcon A (N=254)
IRITIS (Eye disorders) | 0 (0) | 1 (1) — Inflammation of the iris. This was classified as unrelated to the study lens.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: Etafilcon A (N=247) | Test: Galyfilcon A (N=254)
Conjunctivitis (Eye disorders) | 21 (35) | 31 (48) — Includes Bacterial, Viral, Allergic, Contact-lens Papillary, Kerato, and Unspecified Conjunctivitis.
CLPU (Eye disorders) | 2 (2) | 12 (13) — Contact Lens Peripheral Ulcer

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days